CLINICAL TRIAL: NCT05052450
Title: Factors Associated With Mortality, Morbidity and Prognosis in Dementia Patients
Status: Completed | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Neslihan Kayahan, Medical Doctor, Gulhane Training and Research Hospital
Other Study IDs: 2021/290
Record Dates: First submitted 2021-09-08; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Dementia; Dementia, Vascular; Dementia With Lewy Bodies; Dementia of Alzheimer Type; Dementia Frontal; Dementia, Mixed
MeSH Terms: conditions — Dementia; Dementia, Vascular; Lewy Body Disease; Mixed Dementias | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Dementia with Alzheimer: Patients previously diagnosed with Alzheimer disease would be included
  Interventions: Other: Observational
- Dementia with Lewy Body Dementia: Patients previously diagnosed with Lewy Body Dementia would be included
  Interventions: Other: Observational
- Dementia with Fronto-Temporal Dementia: Patients previously diagnosed with Fronto-Temporal Dementia would be included
  Interventions: Other: Observational
- Dementia with Vascular Disease: Patients previously diagnosed with Dementia with Vascular Disease would be included
  Interventions: Other: Observational
- Dementia with Parkinson Disease: Patients previously diagnosed with Dementia with Parkinson Disease would be included
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Patients data were collected throughout the following time

SUMMARY:
Dementia; It is a chronic syndrome characterized by a general and progressive deterioration in cognition, including memory, orientation, language, and comprehension. The prognosis of this progressive and neurodegenerative disease after diagnosis may differ between individuals. In its broadest sense, the prognosis after a diagnosis of dementia; can be defined by shortening of life span, high level of cognitive and functional loss, decrease in quality of life and increased need for care. However, the prognosis of different types of dementia is highly variable. Because it is the most common type of dementia, studies are usually on Alzheimer's disease. It constitutes 50-75% of total dementia cases. Vascular dementia is the second most common cause of dementia and accounts for approximately 15% of dementia cases. Dementia with Lewy bodies constitutes 10-20% of the total dementia patients and ranks second among degenerative dementia types. Frontotemporal dementia, which mimics psychiatric disorders and has prominent behavioural problems, and Parkinson's disease-associated dementia, which is characterized by cognitive impairment that can be added to the existing picture in Parkinson's patients, are also counted among other types of dementia. Prognosis-related data on dementia types other than Alzheimer's disease are limited in the literature. Determining the prognosis is important to support patients, anticipate long-term health problems, plan physician and healthcare provision, and support patients with dementia.In view of the lack of sufficient data on dementia types other than Alzheimer's disease, it is aimed to contribute to the literature on this subject and to determine the factors that may affect prognosis, morbidity and mortality in patients belonging to all dementia types.

ELIGIBILITY:
Inclusion Criteria:

Having applied to the Gulhane Training and Research Hospital Geriatrics Polyclinic Being diagnosed with Alzheimer or Lewy Body Dementia or Vascular Dementia or Fronto-Temporal Dementia or Parkinson Disease Dementia Being at the age of 60 years or older

Exclusion Criteria:

Being under the age of 60 Patients with insufficient recorded data and follow-up for the study Patients who either have diagnosis or follow-up in another center. Patients who have severe dementia that prevents applying for outpatient clinic

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with any kind of dementia and being older than 60 years would be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 2 years
  The event of death occuring during the follow-up period
Mini-Mental State Examination | 2 years
  It was performed to assess mental status. It gives an overall opinion on cognitive domains and tests orientation, registration, attention and calculation, recall, and language. Total scores on Mini-Mental State Examination range from 0 to 30, higher scores show better cognitive performance.
Barthel Index | 2 years
  It was used for assessing physical functioning as a part of the routine geriatric evaluation.where the ten performance items used. Those items defined as feeding, bathing, grooming, dressing, continence of bowel and bladder, toilet use, transfers (bed to chair and back), mobility (on level surfaces), and climbing stairs. Each item is scored on this scale, and the sum is obtained by adding the score of each item (range, 0-100; higher scores show better performance)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naharci MI, Kayahan Satis N, Ozsurekci C, Tasci I. Assessment of clinical features and coexisting geriatric syndromes in newly diagnosed dementia with Lewy bodies: a retrospective study in a tertiary geriatrics setting in Turkey. Eur Geriatr Med. 2023 Feb;14(1):19-27. doi: 10.1007/s41999-022-00727-0. Epub 2022 Dec 13. PMID 36512254